CLINICAL TRIAL: NCT04825184
Title: The Dove Self-Esteem Project: A Randomised Controlled Evaluation Assessing the Impact of a Body Image Chatbot on Brazilian Adolescents' Body Confidence
Brief Title: The Impact of an Artificial Intelligence Chatbot on Brazilian Adolescents' Body Image
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); UNICEF (Other); Talk 2 U (Unknown); Instituto Federal Sudeste de Minas Gerais (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAS.19.12.090
Record Dates: First submitted 2020-11-18; First posted 2021-04-01 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-04

CONDITIONS: Body Image
Keywords: Body image; Adolescents; Brazil; Prevention; Micro-intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blinded to condition allocation (dummy coded) when conducting statistical analyses on primary and secondary trait outcomes; however, blind analyses cannot be conducted on primary and secondary state measures due to the within-group design. Two datasets will be created one for between group analyses with dummy coding, and a second dataset for within group analyses without dummy coding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body image chatbot (Experimental): The artificial intelligence chatbot, Topity, is designed to target sociocultural risk and protective factors for body image using eight therapeutic techniques derived from several evidence-based theories, including media literacy, cognitive behaviour theory and positive body image. The intervention aims to engage users in techniques that teaches users how to 1) Critically analyse and evaluate media content to reduce vulnerability to negative media influences (i.e., media literacy theory; 10); 2) Identify and challenge unhelpful thinking styles and behaviours that perpetuate body image distress (i.e., cognitive behaviour theory; 11); and 3) Appreciating the features, functions and health of the body, beyond it's appearance (i.e., positive body image theory; 12). Users will be assessed on state body satisfaction and affect before and after engaging with a technique to assess the immediate impact of the micro-intervention.
  Interventions: Behavioral: Body image chatbot
- Assessment only (No Intervention): The comparison control condition will be assessment only. This is informed by a care as usual framework; whereby, Brazilian adolescents are not currently offered online body image prevention or intervention resources at school or within the community.

INTERVENTIONS:
Behavioral: Body image chatbot — See arm/group description.
  Other Names: Topity
  Arms: Body image chatbot

SUMMARY:
High prevalence of body and eating concerns in Brazilian populations is well-documented, with risk observed across the lifespan. Prevalence rates of body dissatisfaction range between 26.6 - 56% and 10.7- 36% for adolescent girls and boys, respectively (1, 2, 3). The prevalence of these disordered attitudes and behaviours are mirrored in older populations, and have shown to manifest within family units (6). Further, Brazilian consumer trends reflect these attitudes and behaviours, with it being the leading country in diet pill consumption and aesthetic surgeries, and second in the world for total aesthetic procedures (i.e., surgical and non-surgical), with 2.27 million procedures conducted annually (8).

Despite the scope of body and eating concerns, few evidence-based interventions have been developed and tested for Brazilian populations and even fewer are accessible, scalable or cost-effective. Harnessing technology to deliver evidence-based care is a key focus for researchers. Micro-interventions (brief, low intensity, self-administered interventions), offer an alternative to traditional, intense interventions that may be unsuitable for milder concerns. Body image micro-interventions have proven effective at providing immediate and short-term improvements in body image among women (9). To date, body image micro-interventions have been developed and evaluated among high-income, White, English-speaking samples, with little research exploring how this intervention model may cater to other cultures and countries.

The aim of the present study is to conduct a randomised controlled trial (RCT) to evaluate the immediate and short-term impact of a chatbot on Brazilian adolescents' body image, affect and body image self-efficacy. Primary outcomes include immediate and short-term changes in state- and trait-based body image, respectively. Secondary outcomes include immediate changes in state-based affect and short-term changes in trait affect and body image self-efficacy.

The chatbot intervention is designed to target sociocultural risk and protective factors for body image using eight, brief therapeutic techniques derived from several evidence-based theories, including media literacy, cognitive behaviour theory and positive body image. The chatbot was developed through a collaboration between Dove (Unilever), United Nations Children's Fund (UNICEF), The Centre for Appearance Research, and Talk 2 U.

The comparison control condition will be assessment only. This is informed by a care as usual framework; whereby, Brazilian adolescents are not currently offered body image prevention or intervention resources at school or within the community.

To undertake this project, 2800 adolescent girls and boys will be recruited through an external research agency. Participants will be randomised to either the chatbot or assessment only conditions. Those in the intervention condition, will be encouraged to engage with the chatbot over a 72-hour period, where they will be assessed on state-body satisfaction and affect immediately before and after completing an intervention technique. All participants will be assessed on trait body image, affect and body image self-efficacy at baseline, post-intervention (72-hours) and at one-week and one-month follow-ups. At completion of the one-month follow-up, all participants will receive a debrief form, outlining the study aims and objectives, and additional resources for body and eating concerns. Those in the assessment only condition will be invited to engage with the chatbot; however, their engagement will not be monitored or assessed. Lastly, to compensate participants for their time, they will receive an electronic voucher to the value of approx. US$25 and US$21, for the intervention and control condition, respectively.

DETAILED DESCRIPTION:
Background

High prevalence of body and eating concerns in Brazilian populations is well-documented, with risk observed across the lifespan. With a population of 211 million people, prevalence rates of body dissatisfaction range between 26.6 - 56% and 10.7- 36% for adolescent girls and boys, respectively (1, 2, 3). Equally, an emerging proportion of adolescents report engaging in disordered eating (i.e., binge eating [10.4%], dietary restriction [8.7%]) and weight control behaviours (i.e., vomit and laxative use [.3 - 7.4%]; 4,5). The prevalence of these disordered attitudes and behaviours are mirrored in older populations, and have shown to manifest within family units (6). A meta-analysis into eating disorder prevalence among Brazilian university students (Mage = 21.6 years) reported 14.9% of students met criteria for an eating disorder, with cases highest among nutrition students (7). Meanwhile, Brazilian parents' perceptions of their child's weight during early adolescence (i.e., 11 years), has shown to predict higher weight gain and engagement in weight control behaviours during late-adolescence (i.e., 18 years; 6). Brazilian consumer trends reflect these attitudes and behaviours, with it being the leading country in diet pill consumption and aesthetic surgeries, and second in the world for total aesthetic procedures (i.e., surgical and non-surgical), with 2.27 million procedures conducted annually (8). Despite the scope of body and eating concerns, few evidence-based interventions have been developed and tested for Brazilian populations and even fewer are accessible, scalable or cost-effective.

It is widely accepted among health professionals, policy makers and governments that the global burden of mental health will never be successfully met by extant health professionals and services alone. Further, current intervention modalities (e.g., face-to-face psychotherapy) may be unnecessary or unsuitable for milder concerns, which may be responsive to lower intensity interventions that demand fewer resources. Harnessing technology to deliver evidence-based care is a key focus for researchers. Micro-interventions (brief, low intensity, self-administered interventions), offer an alternative to traditional, intense interventions that may be unsuitable for milder concerns. Body image micro-interventions have proven effective at providing immediate and short-term improvements in body image among women (9). To date, body image micro-interventions have been developed and evaluated among high-income, White, English-speaking samples, with little research exploring how this intervention model may cater to other cultures and countries. Given the prevalence of body image concerns among Brazilian adolescents, coupled with health care disparities, developing evidence-based micro-interventions for scalability is an imperative step in mental health research for Brazil.

The aim of the present study is to evaluate a chatbot that targets risk and protective factors for body image among Brazilian adolescents. Using a two-armed randomised controlled trial design (i.e., intervention vs. assessment only), the study will assess the chatbot's efficacy at eliciting immediate and short-term improvements in adolescents' state- and trait-based body image, affect and body image self-efficacy. This is the first artificial intelligence chatbot to target body image among adolescents, particularly in Brazil; thus, a secondary aim is to assess user's intervention engagement and adherence.

A set of hypotheses were formulated for overall chatbot efficacy (H1-H2), moderation effects within sub-samples (H3) and intervention engagement and adherence (H4):

H1: The chatbot was designed to provide immediate benefits to users. Therefore, it is anticipated that adolescents will experience improvements in state-based body satisfaction and affect at the time of engagement with the chatbot.

H2: Adolescents randomised into the intervention condition will experience greater improvements in trait-based body esteem, affect and body image self-efficacy at post-intervention, one-week and one-month follow-up following a 72-hour trial period, relative to the assessment only control condition.

H3: Intervention effects will be moderated by gender, and baseline levels of body esteem, affect and body image self-efficacy. Specifically, intervention effects will be greatest among:

* Girls
* Girls and boys with lower levels of trait body esteem
* Girls and boys with higher levels of trait negative affect
* Girls and boys with higher levels of body image self-efficacy

H4: With regards to user engagement and adherence, given the novelty of this intervention, analyses will be of an exploratory nature. It is, however, anticipated that greater engagement and adherence with the chatbot intervention will lead to greater improvements in trait-based outcomes.

Design

This is a two-arm randomised controlled trial, comparing an online intervention to an assessment only control condition. Those in the intervention condition will interact with an artificial intelligence chatbot over a 72-hour period, while participants in the control condition will receive care as usual. Assessments of primary and secondary trait outcomes will be conducted at baseline (T1), post-intervention (T2), one-week (T3) and one-month follow-up (T4). Participants in the intervention condition will also be assessed on state body satisfaction and affect immediately before and after engaging with an intervention technique embedded into the chatbot.

Intervention

The body image chatbot, Topity, is designed to target sociocultural risk and protective factors for body image using eight, brief therapeutic techniques derived from several evidence-based theories, including media literacy, cognitive behaviour theory and positive body image. The intervention aims to engage users in techniques that teach users how to 1) Critically analyse and evaluate media content to reduce vulnerability to negative media influences (i.e., media literacy theory; 10); 2) Identify and challenge unhelpful thinking styles and behaviours that perpetuate body image distress (i.e., cognitive behaviour theory; 11); and 3) Appreciating the features, functions and health of the body, beyond it's appearance (i.e., positive body image theory; 12).

Participants

This universal intervention was designed to provide whole population benefits, irrespective of an individual's level of risk. Therefore, increased risk for body or eating concerns was not an inclusion criterion for this trial. Eligible participants are those aged 13-18 years old; Portuguese speaking; Brazilian resident; and, have access to Facebook Messenger.

Recruitment and data collection procedures

A representative sample of 2,800 adolescents aged 13-18 will be recruited via a Brazilian research agency, using the agency's recruitment panels (e.g., via email) and UNICEF's online communication platforms (e.g., U-Report). Recruitment materials will include a link to a screener to determine participant eligibility.

Based on the screening results, participants will receive an information pack to be read by themselves and their parent or guardian. Parents will be invited to provide consent by uploading a signed consent to an online, confidential portal. Following parent consent, participants will complete the online self-report assessment (baseline; T1), which will commence with adolescents providing informed assent, by clicking a checkbox. Those who do no assent will not proceed with the trial. At completion of the baseline survey, adolescents will be randomised into one of two conditions: intervention or assessment only. Those in the intervention condition will receive a link to the chatbot via email 24-hours after completing the baseline assessment. Those in the assessment only condition will be advised of their opportunity to engage with the chatbot at study completion.

Adolescents will be invited and encouraged to engage with the chatbot, as much as possible, over a 72-hour period. During this period, participants will have the opportunity to complete and re-engage with eight intervention techniques. Participants will be assessed on state body satisfaction and affect immediately after engaging with a technique. At the completion of the 72-hour period, both conditions will be assessed on primary and secondary trait outcomes (post-intervention; T2). Those in the intervention condition will be encouraged to continue using the chatbot. One-week (T3) and one-month (T4) following the intervention period, participants will be assessed on primary and secondary trait outcomes. At the completion of the one-month follow-up, all participants will receive a debrief form, outlining the study aims and objectives, and additional resources for body image and eating concerns. Those in the assessment only condition will be invited to engage with the chatbot; however, their engagement will not be monitored or assessed.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 13-18 years old; Portuguese speaking; Brazilian resident; and, have access to Facebook Messenger.

Exclusion Criteria:

* N/A

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1715 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Change in state body satisfaction | Immediately pre-intervention and immediately post-intervention (change)
  Measured via a 11-point Likert scale (0 = not at all satisfied; 10 = very satisfied).
Change in trait body image | Baseline, post-intervention (72-hours following baseline assessment), one-week follow-up (7-days following post-intervention assessment) and one-month follow-up (28-days following post-intervention assessment).
  Brazilian version of the Body Esteem Scale for Adolescents and Adults (BESAA; 13); a 23-item scale, comprising of three subscales: appearance esteem, weight esteem and attribution. Responses are scored on a 5-point Likert scale (1 = never to 5 = always).

SECONDARY OUTCOMES:
Change in state affect | Immediately pre-intervention and immediately post-intervention (change)
  Measured via a 11-point Likert scale (0 = not at all happy; 10 = very happy).
Change in trait affect | Baseline, post-intervention (72-hours following baseline assessment), one-week follow-up (7-days following post-intervention assessment) and one-month follow-up (28-days following post-intervention assessment).
  Brazilian version of the Positive and Negative Affect Scale for Children (PANAS-C8; 14); eight words related to positive (e.g., joyful) and negative (e.g., irritated) emotive states. Responses are score on a 5-point Likert scale (1 = not at all to 5 = extremely); participants indicate the degree to which they have experienced the emotion in a preceding time-frame.
Change in body image self-efficacy | Baseline, post-intervention (72-hours following baseline assessment), one-week follow-up (7-days following post-intervention assessment) and one-month follow-up (28-days following post-intervention assessment).
  Developed by the authors according to Bandura's guidelines for constructing self-efficacy questionnaires. Items were informed by self-efficacy scales developed specifically for depression (15) and diabetes (16); 5-item scale assesses participants' beliefs in their ability to execute behaviours that manage body image distress. Items are scored on a 101-point Visual Analogue Scale (VAS), ranging from 0 (i.e., 'not at all confident') to 100 (i.e., 'very confident').
Total acceptability of the intervention | Through intervention completion, over the course of 72-hours.]
  Acceptability of the intervention will be assessed at completion of the 72-hour trial period using nine 101-point Visual Analogue Scales. The nine items assess the participants perception of the chatbot, including level of interestedness, enjoyment, relevance, helpfulness, likelihood to recommend and re-engage, and ease of engagement (i.e., level of ease, speed, accuracy). An acceptability mean score will be created from the nine items.
Total intervention adherence | Through intervention completion, over the course of 72-hours.
  Participants need to complete a minimum of one intervention technique over the course of the 72-hour intervention period. Completion will be coded as 1, with non-completion coded as 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Toluna, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amaral ACS, Stice E, Ferreira MEC. A controlled trial of a dissonance-based eating disorders prevention program with Brazilian girls. Psicol Reflex Crit. 2019 Jun 17;32(1):13. doi: 10.1186/s41155-019-0126-3. PMID 32026167
- [Background] Moehlecke M, Blume CA, Cureau FV, Kieling C, Schaan BD. Self-perceived body image, dissatisfaction with body weight and nutritional status of Brazilian adolescents: a nationwide study. J Pediatr (Rio J). 2020 Jan-Feb;96(1):76-83. doi: 10.1016/j.jped.2018.07.006. Epub 2018 Aug 9. PMID 30098939
- [Background] Santana ML, Silva Rde C, Assis AM, Raich RM, Machado ME, de J Pinto E, de Moraes LT, Ribeiro Junior Hda C. Factors associated with body image dissatisfaction among adolescents in public schools students in Salvador, Brazil. Nutr Hosp. 2013 May-Jun;28(3):747-55. doi: 10.3305/nh.2013.28.3.6281. PMID 23848099
- [Background] Leal GVDS, Philippi ST, Alvarenga MDS. Unhealthy weight control behaviors, disordered eating, and body image dissatisfaction in adolescents from Sao Paulo, Brazil. Braz J Psychiatry. 2020;42(3):264-270. doi: 10.1590/1516-4446-2019-0437. Epub 2020 Jan 31. PMID 32022158
- [Background] Silva SUD, Barufaldi LA, Andrade SSCA, Santos MAS, Claro RM. Nutritional status, body image, and their association with extreme weight control behaviors among Brazilian adolescents, National Adolescent Student Health Survey 2015. Rev Bras Epidemiol. 2018 Nov 29;21(suppl 1):e180011. doi: 10.1590/1980-549720180011.supl.1. English, Portuguese. PMID 30517462
- [Background] Abdalla S, Buffarini R, Weber AM, Cislaghi B, Costa JC, Menezes AMB, Goncalves H, Wehrmeister FC, Meausoone V, Victora CG, Darmstadt GL. Parent-Related Normative Perceptions of Adolescents and Later Weight Control Behavior: Longitudinal Analysis of Cohort Data From Brazil. J Adolesc Health. 2020 Jan;66(1S):S9-S16. doi: 10.1016/j.jadohealth.2019.09.007. PMID 31866039
- [Background] Trindade AP, Appolinario JC, Mattos P, Treasure J, Nazar BP. Eating disorder symptoms in Brazilian university students: a systematic review and meta-analysis. Braz J Psychiatry. 2019 Mar-Apr;41(2):179-187. doi: 10.1590/1516-4446-2018-0014. Epub 2018 Oct 11. PMID 30328965
- [Background] International Association for Aesthetic/Cosmetic Surgery. (2017). ISAPS International Survey on Aesthetic/Cosmetic Procedures Performed in 2017. ISAPS. https://www.isaps.org/wpcontent/uploads/2019/03/ISAPS_2017_International_Study_Cosmetic_Procedures_NEW.pdf
- [Background] Fuller-Tyszkiewicz, M., Richardson, B., Lewis, V., Linardon, J., Mills, J., Juknaitis, K., ... & Ware, A. (2019). A randomized trial exploring mindfulness and gratitude exercises as eHealth-based micro-interventions for improving body satisfaction. Computers in Human Behavior, 95, 58-65.
- [Background] Aufderheide, P. (1993). Media Literacy. A Report of the National Leadership Conference on Media Literacy. Aspen Institute, Communications and Society Program, 1755 Massachusetts Avenue, NW, Suite 501, Washington, DC 20036.7
- [Background] Cash, T. F. (2002). Body image: Cognitive behavioral perspectives on body image. Body images: A handbook of theory, research, and clinical practice, 38-46.
- [Background] Menzel, J. E., & Levine, M. P. (2011). Embodying experiences and the promotion of positive body image: The example of competitive athletics.
- [Background] Mendelson BK, Mendelson MJ, White DR. Body-esteem scale for adolescents and adults. J Pers Assess. 2001 Feb;76(1):90-106. doi: 10.1207/S15327752JPA7601_6. PMID 11206302
- [Background] Damásio, B. F., Pacico, J. C., Poletto, M., & Koller, S. H. (2013). Refinement and psychometric properties of the eight-item Brazilian positive and negative affective schedule for children (PANAS-C8). Journal of Happiness Studies, 14(4), 1363-1378.
- [Background] Bandura, A. (1982). Self-efficacy mechanism in human agency. American psychologist, 37(2), 122.
- [Background] McCusker J, Lambert SD, Cole MG, Ciampi A, Strumpf E, Freeman EE, Belzile E. Activation and Self-Efficacy in a Randomized Trial of a Depression Self-Care Intervention. Health Educ Behav. 2016 Dec;43(6):716-725. doi: 10.1177/1090198116637601. Epub 2016 May 13. PMID 27179288
- [Background] Williams GC, Freedman ZR, Deci EL. Supporting autonomy to motivate patients with diabetes for glucose control. Diabetes Care. 1998 Oct;21(10):1644-51. doi: 10.2337/diacare.21.10.1644. PMID 9773724
- [Derived] Matheson EL, Smith HG, Amaral ACS, Meireles JFF, Almeida MC, Linardon J, Fuller-Tyszkiewicz M, Diedrichs PC. Using Chatbot Technology to Improve Brazilian Adolescents' Body Image and Mental Health at Scale: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Jun 19;11:e39934. doi: 10.2196/39934. PMID 37335604
- [Derived] Matheson EL, Smith HG, Amaral ACS, Meireles JFF, Almeida MC, Mora G, Leon C, Gertner G, Ferrario N, Suarez Battan L, Linardon J, Fuller-Tyszkiewicz M, Diedrichs PC. Improving body image at scale among Brazilian adolescents: study protocol for the co-creation and randomised trial evaluation of a chatbot intervention. BMC Public Health. 2021 Nov 20;21(1):2135. doi: 10.1186/s12889-021-12129-1. PMID 34801002